CLINICAL TRIAL: NCT04542655
Title: An Open-label, Single-center, Randomized, Controlled, Exploratory Study to Investigate the Effect of Weight Bearing Versus Non-weight Bearing Exercise on Collagen and Proteoglycan in Serum and Urine in Patients With Osteoarthritis and Healthy Subjects
Brief Title: The Effect of Exercise on Serum Levels of Collagen and Proteoglycan in Patients With Knee Osteoarthritis (EFEX-OA-01)
Acronym: EFEX-OA-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Bioscience A/S (Industry)
Collaborators: University of Copenhagen (Other); NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EFEX-OA_Protocol_Final_v1.1
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to an order of exercise-intervention: cycling, running. This will be followed by a resting intervention. Interventions are planned 1 week apart.
  Blood will be sampled before, immediately after and again at 1, 2, 3 and 24 hours after intervention start. Spot urine is sampled before, after and the next day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycling first (Other): Ergometer cycling then treadmill running then rest
  Interventions: Other: Ergometer Cycling followed by treadmill running; Other: Rest
- Running first (Other): Treadmill running then ergometer cycling then rest
  Interventions: Other: Treadmill Running followed by ergometer cycling; Other: Rest

INTERVENTIONS:
Other: Ergometer Cycling followed by treadmill running — The participants undergo ergometer cycling, treadmill running and rest.
  Other Names: Exercise
  Arms: Cycling first
Other: Treadmill Running followed by ergometer cycling — The participants undergo treadmill running, ergometer cycling and rest.
  Other Names: Exercise
  Arms: Running first
Other: Rest — The participants undergo ergometer cycling, treadmill running and rest.
  Other Names: Non Exercise

SUMMARY:
Aim of EFEX-OA-01: To explore how running, cycling and resting acutely influence levels of collagen and proteoglycan in patients with osteoarthritis knee and in young healthy subjects, as reflected by changes in serum and urine biochemical markers originating from joint related collagens and proteoglycans.

ELIGIBILITY:
Inclusion criteria for OA patients:

1. Kellgren-Lawrence radiological grade of 1-3 in at least one tibio-femoral joint diagnosed by screening x-ray.
2. 35 to < 75 years of age at the time of signing the informed consent form.
3. Bodyweight > 50 and < 150 kg and a BMI in the range 18,5-35 kg/m2.
4. Are male or female.
5. Is able to meet for all of the four study visits and comply with the dietary and activity restrictions.
6. Can give informed consent.

Exclusion criteria for OA patients:

Medical conditions:

1. History of arthroscopy or intra-articular administration of corticosteroids or hyaluronic acid into the target knee within 6 months before screening.
2. Kellgren-Lawrence radiological grade of 4 in at least one tibio-femoral joint
3. Previous arthroplasty of knee or hip.
4. Intention of having major surgery during the timeframe of this study.
5. OA related to eg. dysplasia, aseptic osteonecrosis, acromegaly, Paget disease, Stickler syndrome, hemochromatosis, gout, chondrocalcinosis (pseudogout) or calcium pyrophosphate deposition disease.
6. Current treatment with beta-receptor adrenergic antagonists (beta-blockers), systemic corticosteroid treatment in doses equivalent to > 10 mg of prednisolone per day, or Vitamin K antagonists, new oral anticoagulants, fractionated and non-fractionated heparin
7. Active systemic infection.
8. Active systemic inflammatory or autoimmune disease.
9. Symptomatic occlusive arterial disease e.g. claudication intermittens.
10. Heart failure > NYHA class II.
11. History of transient ischaemic attack or stroke.
12. ECG findings which, in the opinion of the investigator, compromises patient safety related to HRmax-test.
13. History of coronary artery disease, myocardial infarction, or other serious cardiovascular disease, as evaluated by the investigator.
14. Is not currently active athlete or a highly trained individual.

Inclusion criteria for healthy subjects:

1. 18 to < 75 years of age at the time of signing the informed consent form.
2. Have a bodyweight within > 50 and < 150 kg and a BMI within the range 18,5-35 kg/m2.
3. Are male or female.
4. Is able to meet for all of the four study visits and comply with the dietary and activity restrictions.
5. Can give informed consent.

Exclusion criteria for healthy subjects:

1. History of arthroscopy or intra-articular administration of corticosteroids or hyaluronic acid into the target knee within 6 months before screening.
2. Previous arthroplasty of knee or hip.
3. Intention of having major surgery during the timeframe of this study.
4. Secondary OA e.g. because of dysplasia, aseptic osteonecrosis, acromegaly, Paget disease, Stickler syndrome, hemochromatosis, gout, chondrocalcinosis (pseudogout) or calcium pyrophosphate deposition disease.
5. Current treatment with beta-receptor adrenergic antagonists (beta-blockers), systemic corticosteroid treatment in doses equivalent to > 10 mg of prednisolone per day, or Vitamin K antagonists, new oral anticoagulants, fractionated and non-fractionated heparin
6. Any known active systemic infection.
7. Any known active systemic inflammatory or autoimmune disease.
8. Symptomatic occlusive arterial disease e.g. Inermittent claudication.
9. Heart failure > NYHA class II.
10. History of transient ischaemic attack or stroke.
11. History of coronary artery disease, myocardial infarction, or other serious cardiovascular disease, as evaluated by the investigator.
12. ECG findings which, in the opinion of the investigator, compromises patient safety related to HRmax-test.
13. Is not currently active athlete or a highly trained individual.
14. X-ray verified Kellgren-Lawrence grade 1-4.
15. Is clinically suspected of having hip OA.

Other exclusions (all subjects):

1. Legal incapacity or limited legal capacity
2. Inability to communicate or cooperate with the investigator or to comply with the requirements of the entire study.
3. Are categorized as being very difficult to draw blood from, as evaluated by the investigator.
4. Current alcohol abuse and/or inability to refrain from intake of alcoholic beverages 24 hours prior to study intervention.
5. Other factors e.g. self-reported drug abuse, which in the opinion of the investigator may interfere with the study conduct.
6. Site staff, study staff members and study staff family members.
7. Other concomitant disease compromising or otherwise significantly affecting ECM turnover in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Changes in biomarkers (exploratory) | Acute: 0-4 hours and subacute: 24 hours
  Serum and urine biochemical markers of collagen and proteoglycan turnover

CONTACTS AND LOCATIONS:
Overall Officials: Henning Nielsen, MD, DMSci, Principal Investigator — Sanos Clinic
Locations (1):
- Sanos Clinic, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjerre-Bastos JJ, Nielsen HB, Andersen JR, Karsdal M, Boesen M, Mackey AL, Byrjalsen I, Thudium CS, Bihlet AR. A biomarker perspective on the acute effect of exercise with and without impact on joint tissue turnover: an exploratory randomized cross-over study. Eur J Appl Physiol. 2021 Oct;121(10):2799-2809. doi: 10.1007/s00421-021-04751-z. Epub 2021 Jun 22. PMID 34156534